CLINICAL TRIAL: NCT01191710
Title: Is the Clinical Outcome Affected by the Incidence of Progesterone Elevation on the Day of hCG Triggering When Agonist Protocol is Compared to Antagonist Protocol for IVF
Brief Title: Progesterone Rise in Agonist Versus Antagonist in Vitro Fertilization (IVF) Cycles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: BioGenesis (Industry)
Responsible Party: Papanikolaou Evangelos, Human Reproduction and Genetics Foundation (HRG)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ProgRise001
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2009-01

CONDITIONS: Pregnancy Outcome After In Vitro Fertilization (IVF)
Keywords: progesterone
MeSH Terms: interventions — Fertilization in Vitro; Pregnancy; Embryo Transfer; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antagonist group (Experimental): Antagonist protocol for IVF
  Interventions: Other: In vitro fertilization
- Agonist group (Active Comparator): Long Agonist protocol for IVF
  Interventions: Other: In vitro fertilization

INTERVENTIONS:
Other: In vitro fertilization — In vitro fertilization procedure with gonadotropin induced follicular ovarian stimulation
  Other Names: IVF; pregnancy; embryo-transfer; progesterone

SUMMARY:
The aim is to explore whether the incidence of progesterone rise in the late follicular phase differs between GnRH-agonist and GnRH-antagonist protocols for IVF and whether this has an impact on the probability of pregnancy achievement.

DETAILED DESCRIPTION:
In view of the current debate concerning possible differences in efficacy between the two GnRH analogues, the current study aimed to explore whether progesterone control in the late follicular phase differs when GnRH-agonist is used as compared to GnRH-antagonist and if so to what extend does the progesterone rise have an impact on the probability of achieving a pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* age < 39
* follicle-stimulating hormone (FSH) < 12
* gonadotropin dose 100-300IU

Exclusion Criteria:

* endometriosis
* known endocrine disorder
* blood analyzed in another laboratory

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of late progesterone rise on the day of HCG triggering | Up to delivery (2010)

SECONDARY OUTCOMES:
Clinical pregnancy rate Delivery rate | Up to delivery (2010)

CONTACTS AND LOCATIONS:
Overall Officials: Basil Tarlatzis, MD, Study Chair — BioGenesis
Locations (1):
- Biogenesis, Thessaloniki, Pylaia, Greece

REFERENCES:
- [Background] Papanikolaou EG, Kolibianakis EM, Pozzobon C, Tank P, Tournaye H, Bourgain C, Van Steirteghem A, Devroey P. Progesterone rise on the day of human chorionic gonadotropin administration impairs pregnancy outcome in day 3 single-embryo transfer, while has no effect on day 5 single blastocyst transfer. Fertil Steril. 2009 Mar;91(3):949-52. doi: 10.1016/j.fertnstert.2006.12.064. Epub 2007 Jun 6. PMID 17555751
- [Derived] Papanikolaou EG, Pados G, Grimbizis G, Bili E, Kyriazi L, Polyzos NP, Humaidan P, Tournaye H, Tarlatzis B. GnRH-agonist versus GnRH-antagonist IVF cycles: is the reproductive outcome affected by the incidence of progesterone elevation on the day of HCG triggering? A randomized prospective study. Hum Reprod. 2012 Jun;27(6):1822-8. doi: 10.1093/humrep/des066. Epub 2012 Mar 14. PMID 22422777
- See also: Related Info — http://www.hrg.gr